CLINICAL TRIAL: NCT04149951
Title: Randomized, Double Blind Controlled Trial to Evaluate Efficacy of Vestibular Nerve Stimulation (VeNS), With Lifestyle Modification, Compared to Control and Lifestyle Modification, as a Means of Lowering HbA1c in Adults With Type 2 Diabetes
Brief Title: Effect of VeSTAL Device in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: Compliance Solutions Ltd. (Industry); University College Dublin (Other); Exploristics Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCD2
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment in 1:1 active to control allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Randomized to active device use plus lifestyle modification (500kcal deficit hypocaloric diet and 150 min of exercise per week for each subject).
  Interventions: Device: Vestal Device
- Control (Placebo Comparator): Randomized to sham device use plus lifestyle modification (500kcal deficit hypocaloric diet and 150 min of exercise per week for each subject).
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: Vestal Device — Vestibular nerve stimulator
  Arms: Active
Device: Placebo device — Sham nerve stimulator
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS), together with a lifestyle modification program, as a method of reducing HbA1c, as compared to a sham control with both study arms incorporating a lifestyle modification program.

* Allocation: Randomized
* Endpoint classification: Efficacy Study
* Intervention Model: Parallel Assignment in 1:1 active to control allocation

DETAILED DESCRIPTION:
There is an ongoing and worsening problem with type 2 diabetes mellitus (DM) in the developed, and much of the developing world. Although it has long been realized that Western diets that are rich in sugar and fat play an important role in this, it has only recently been realized that exposure to these diets, particularly in childhood, can damage the part of the brain that determines how much fat there is in the body, which may well play a role in the development of metabolic syndrome, deranged glycemic control and type 2 DM. It is believed, based on animal and human work, that VeNS pushes the set-point for fat downwards to cause fat loss, possibly because this indicates to the brain a state of increased physical activity. VeNS may additionally have other direct, yet to be quantified, effects on glycemic control.

The sponsors have unpublished pilot data from Dr Saisailesh Kumar at RDG Medical College in India that show an improvement in glycemic control can be achieved by one hour a day of VeNS over a three month period. Both groups received a hypocaloric diet tailored to diabetics. The aim of this study is to determine whether this effect can be replicated in a slightly larger European based population.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 DM
2. HbA1c ≥7.0% and ≤10.0%
3. If on oral anti-diabetic medication should be stable dosage regime last 3 months
4. Males or Females. Note females of child-bearing potential must have a negative urine pregnancy test.
5. 18-80 years of age inclusive on starting the study.
6. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with: trying to use the device on a daily basis; the hypocaloric diet weight loss program; and this provided weight loss support and mentoring.
7. Agreement not to use of prescription, or over-the-counter, weight loss preparations for the duration of the trial.
8. Agreement not to start smoking tobacco or marijuana for the duration of the study.
9. Access to Wi-Fi (to connect iPod to internet)

Exclusion Criteria:

1. History of vestibular dysfunction or other inner ear disease as indicated by the screening questions.
2. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
3. History of weight loss device implantation (e.g. VBloc Maestro or Abiliti).
4. Use of a non-invasive weight loss device (e.g. Modius)
5. Hypothyroidism requiring current treatment with levothyroxine (e.g. Levo-T, Synthroid, Thyroxine) (Other thyroid disorder patients on stable treatment for at least 3 months are acceptable).
6. Other endocrinological causes of weight gain (e.g. Cushing's disease, Cushing's syndrome or acromegaly)
7. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working).
8. Diagnosis of liver, kidney or heart failure.
9. Tobacco or marijuana smoking in the 3 months before starting and for the duration of the study.
10. Known genetic cause of type 2 DM (e.g., Prader-Willi Syndrome).
11. Current, active member of an organized weight loss program.
12. Diagnosis of Type 1 DM.
13. Use of insulin.
14. Diagnosis of epilepsy or use of anti-epileptic medication within 3 months of starting the study (e.g. for the treatment of peripheral neuropathy)
15. Use of oral or intravenous corticosteroid medication within 3 months of starting the study.
16. Use of the beta-blockers within 3 months of starting the study.
17. Current alterations in treatment regimens of anti-depressant medication for whatever reason (including tricyclic antidepressants) (Note: stable treatment regimen for prior 6 months acceptable).
18. A myocardial infarction within the preceding year.
19. A history of stroke or severe head injury (as defined by a head injury that required craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).
20. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
21. Untreated severe depression, schizophrenia, substance abuse, and eating disorder.
22. Current participant in another clinical trial.
23. Have a family member who is currently participating or is planning to participate in this study.
24. Pregnancy.
25. Blood transfusion within 4 months, or need for recurrent transfusions.
26. Hemolytic anemias including sickle cell, thalassemia and autoimmune varieties.
27. Hemochromatosis.
28. Use of dietary/ herbal supplements to assist with diabetic control.
29. History of migraine headaches.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | 4 months
  Percentage

SECONDARY OUTCOMES:
Difference in mean weight loss between the active-product and sham-treated groups. | 4 months
  Grams
Daily caloric intake | 4 months
  Two day 24 hour recall
Blood pressure | 4 months
  mmHg
Waist circumference | 4 months
  cm
Hip circumference | 4 months
  cm
Body mass index | 4 months
  kg/m2
Appetite | 4 months
  Rating from -1 to 1
Cravings | 4 months
  Rating from -1 to 1
Fullness | 4 months
  Rating from -1 to 1

OTHER OUTCOMES:
Mentorship support usage | 4 months
  Average hours per week
Dose response analysis | 4 months
  Average hours per week

CONTACTS AND LOCATIONS:
Overall Officials: Carel Le Roux, MD PhD, Principal Investigator — UCD
Locations (1):
- St Vincents Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No